CLINICAL TRIAL: NCT05519202
Title: A Single-arm, Single-center Exploratory Clinical Study of Penpulimab Injection Combined With SOX in the Perioperative Treatment of Gastric Cancer
Brief Title: Exploratory Clinical Study of Penpulimab Combined With SOX in the Perioperative Treatment of Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJLS-KLDMIR-22209
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer, SOX, PD-1, perioperative period
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SOX and Penpulimab (Experimental): S-1 ( 40 mg/m2 bid po d1-14) and Penpulimab (200mg ivgtt d1) and Oxaliplatin ( 130 mg/m2 (d1) The treatment period of the above drugs was 3 weeks, and the duration of preoperative treatment was 3 cycles. After treatment, the patient underwent surgery after evaluation. Four cycles of adjuvant therapy with the original regimen (preoperative) were performed after surgery.
  Interventions: Drug: S-1,Oxaliplatin, Penpulimab

INTERVENTIONS:
Drug: S-1,Oxaliplatin, Penpulimab — S-1 ( 40 mg/m2 bid po d1-14) and Penpulimab (200mg ivgtt d1) and Oxaliplatin ( 130 mg/m2 (d1)
  Other Names: SOX and Penpulimab

SUMMARY:
To explore the efficacy and safety of Penpulimab combined with SOX in the perioperative treatment of gastric cancer

DETAILED DESCRIPTION:
Gastric cancer is one of the malignant tumors that seriously threaten human health. It is the sixth most common malignant tumor in the world. According to Global Cancer Statistics 2020, there were about 1.089 million new cases of gastric cancer and 768,000 deaths of gastric cancer worldwide in 2020. Multidisciplinary treatment with radical surgical resection as the core is the mainstream mode of comprehensive treatment of gastric cancer at present, and radical gastrectomy is recognized as the best treatment. However, for patients with advanced gastric cancer, the effect of surgery alone is not good, and the postoperative tumor recurrence rate is high. In order to improve the disease-free survival rate and overall Surv Ival (OS) rate of gastric cancer patients after surgery, perioperative comprehensive therapy has been gradually adopted by the majority of scholars, and has achieved encouraging efficacy in clinical application.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent;
* At least 18 years of age;
* ECOG PS: 0-1;
* Patients with gastric cancer diagnosed as T3-4NXMX by imaging;
* Patients with gastric adenocarcinoma diagnosed by cytology;
* Patients with gastric cancer assessed by the surgeon as suitable for neoadjuvant therapy or conversion therapy followed by radical resection;
* Laboratory tests should meet the following requirements (28 days before enrollment in baseline period) :
* Women should agree that they must use contraception during and for 6 months after the study; Had a negative serum pregnancy test within 7 days prior to study enrollment and had to be non-lactating; Men should agree that they must use contraception during the study and for 6 months after the end of the study period.

Exclusion Criteria:

* Co-existing with other malignant tumors (except cured basal cell carcinoma of the skin);
* Gastric cancer patients with T1-2N0M0;
* Previous treatment including anti-PD-1 /PD-L1/CTLA-4 antibody therapy or other immunotherapy directed against PD-1/PD-L1/CTLA-4;
* Weight loss greater than or equal to 20% within 4 weeks before the first dose;
* Severe hypersensitivity after administration of other monoclonal antibodies;
* The presence or history of any active autoimmune disease
* Immunosuppressive therapy, systemic or absorbable local hormone therapy (dose > 10mg/ day prednisone or other effective hormone) is required to achieve immunosuppression and continues to be used within 2 weeks of the first administration;
* Patients with multiple factors affecting oral medication
* Uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage;
* Had received a prophylactic or attenuated vaccine within 4 weeks before the first dose;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response(pCR) | 2 years
  the proportion of patients got pathological complete response rate

SECONDARY OUTCOMES:
The 1-year DFS rate | 1 years
  the proportion of patients without relapse
The 1-year OS rate | 1 years
  OS was defined as the time from first day of study treatment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up
Disease free survival,DFS | 2 years
  defined as, according to the RECIST1.1 criteria, the time between subjects from enrollment to disease recurrence or death (for any reason)
Overall Response Rate (ORR) | 2 years
  ORR was defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1
tumor regression grade(TRG) | 2 years
  Ryan's 0-3 classification method was used